CLINICAL TRIAL: NCT06755684
Title: Neoadjuvant Befotertinib Combined Bevacizumab or Platinum-based Double Chemotherapy for Resectable Locally-advanced EGFR Mutation-positive Non-Small Cell Lung Cancer: a Single-center, Randomized Controlled Trial
Brief Title: Neoadjuvant Befotertinib Combined Bevacizumab or Platinum-based Double Chemotherapy for Resectable Locally-advanced EGFR Mutation-positive Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peng Zhang (Other)
Responsible Party: Sponsor-Investigator, Peng Zhang, Archiater, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-021
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: EGFR; Non-Small Cell Lung Cancer; Locally Advanced Non-Small Cell Lung Cancer; Pemetrexed; Carboplatin; Bevacizumab; Antineoplastic Agents; Tyrosine Kinase Inhibitor
Keywords: EGFR-TKI; NSCLC; Chemotherapy; Bevacizumab; Locally advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Befotertinib combined Bevacizumab (Experimental): Befotertinib combined Bevacizumab
  Interventions: Drug: Befotertinib combined Bevacizumab
- Befotertinib combined platinum-based double chemotherapy (Experimental): Befotertinib combined platinum-based double chemotherapy
  Interventions: Drug: Befotertinib combined platinum-based double chemotherapy

INTERVENTIONS:
Drug: Befotertinib combined Bevacizumab — Befotertinib combined Bevacizumab
  Arms: Befotertinib combined Bevacizumab
Drug: Befotertinib combined platinum-based double chemotherapy — Befotertinib combined platinum-based double chemotherapy
  Arms: Befotertinib combined platinum-based double chemotherapy

SUMMARY:
This study targeted patients with resectable stage II-IIIA non-small cell lung cancer with EGFR mutation

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patient with EGFR sensitive mutation as confirmed by needle biopsy;
* At stage II-IIIA (TNM Staging, Version 8) as identified by chest CT, PET-CT or/and EBUS;
* No systemic metastasis (confirmed by head MRI, whole body bone scan, PET-CT, liver and adrenal CT, etc.);
* With the feasibility to receive radical surgery ;
* Good lung function that could tolerate surgical treatment;
* Aged 18-75 years;
* At least one measurable tumor foci (the longest diameter measured by CT shall be > 10 mm);
* Other major organs shall function well (liver, kidney, blood system, etc.):
* ECOG PS score shall be 0-1;
* The child-bearing female must undergo pregnancy test within 7 days before starting the treatment and the result shall be negative. Reliable contraceptive measures, such as intrauterine device, contraceptive pill and condom, shall be adopted during the trial and within 30 days after completion of the trial. The child-bearing male shall use condom for contraception during the trial and within 30 days after completion of the trial;
* The patient shall sign the Informed Consent Form.

Exclusion Criteria:

* The patient has undergone any systemic anti-cancer treatment for NSCLC, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment, etc.;
* The patient suffers from any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina pectoris, angina pectoris that starts to attack within the last 3 months, congestive heart failure [≥ Grade II specified by New York Heart Association (NYHA)], cardiac infarction (6 months before enrollment), severe arrhythmia and liver, kidney or metabolic diseases that requires drug treatment;
* The patient is a carrier of HIV;
* The patient has had or is currently suffering from interstitial lung disease;
* The patient had undergone other major systemic operations or suffered from severe trauma within 3 months before the trial;
* The patient is allergic to befotertinib or its any excipients;
* The patient is allergic to bevacizumab or its any excipients;
* The patient is allergic to platinum-based double chemotherapy or its any excipients;
* The female patient is in pregnancy or lactation period;
* There are any conditions under which the investigator considers the patient is not suitable to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | up to 4 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 4 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy. Only patients with measurable lesions at baseline will be analyzed.
Progression-free survival (PFS) | up to 60 months
  It refers to the time (months) from the first administration of drug in this study to the disease progression or death (including any cause of death in the case of no progression) as recorded in CRF, regardless of whether the patient exits from the treatment or receives other anti-cancer treatment before progression.
Event-free survival (EFS) | Up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Disease-free survival (DFS) | up to 60 months
  It refers to the time (months) from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
R0 rate | up to 4 months
  It is defined as the rate of complete resection with no residual tumor cell in the resection margin.
adverse event (AE) rate | up to 4 months
  It is defined as the frequency of adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.
Complete Pathological response (CPR) | Up to 4 months
  CPR is defined as the proportion of participants who have achieved complete pathologic response (on routine hematoxylin and eosin staining, tumors with no viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided